CLINICAL TRIAL: NCT05755009
Title: High- and Low-dose Radiotherapy Combined With Envafolimab for Metastatic Solid Tumor: A Single-arm, Single-center, Phase II Trial
Brief Title: High- and Low-dose Radiotherapy Combined With Envafolimab for Metastatic Solid Tumor
Acronym: ST-CR01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Solid tumor-CR01
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Cancer
Keywords: Metastatic solid tumor; immune checkpoint inhibitors; radiotherapy; Objective response rate
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High- and Low-dose radiotherapy combined with immunotherapy (Experimental): High- and Low-dose radiotherapy combined with immunotherapy and maintain immunotherapy. Immunotherapy (Envafolimab) once every week (maintain total two years). Continuous high-(8Gy×5F) and low-dose (1.33Gy×5F) Radiotherapy starts at the second week after immunotherapy.
  Interventions: Radiation: High- and Low-dose radiotherapy

INTERVENTIONS:
Radiation: High- and Low-dose radiotherapy — High- and Low-dose radiotherapy combined with immunotherapy and maintain immunotherapy. Immunotherapy (Envafolimab) once every week (maintain a total of two years). Continuous high-(8Gy×5F) and low-dose (1.33Gy×5F) Radiotherapy starts at the second week after immunotherapy.

SUMMARY:
The purpose of this study is to explore the efficacy and safety of high- and low-dose radiotherapy (HD-RT/LD-RT) combined with envafolimab (I) in the treatment of metastatic solid tumors that have failed first-line immunotherapy or above.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastasis (including recurrence) solid tumors and failure with first-line or above immunotherapy (PD-1/PD-L1/CTLA-4 inhibitors), and no subsequent standard treatment regimen.
2. Previous histopathologic confirmation of malignancy.
3. Tumor diameter > 5 cm or the number of metastases is 6-15 (at least one measurable lesion, bone metastases are not used as target lesions), not suitable for conventional radiotherapy, surgery, radiofrequency ablation, and other treatments.
4. Patients with an ECOG score of 0 or 1, and an expected survival period of ≥6 months.
5. During the study, they are willing to follow the arrangement and not use other systemic anti-tumor drugs such as chemotherapy, targeted, Chinese herbal medicine, and proprietary Chinese medicine.
6. 18-70 years old, no gender limit.

Exclusion Criteria:

* 1. Patients with glioma or brain metastases. 2. Those with a history of severe immediate allergy to the drugs used in this study.

  3. Suffered from other malignant tumors other than nasopharyngeal carcinoma within 5 years (except for tumors with an expected 5-year OS>90%, such as non-melanoma skin cancer or pre-invasive cervical cancer).

  4. Cancer patients who require urgent surgical intervention, such as high-risk pathological fractures, life-threatening bleeding symptoms, etc.

  5. Any of the following conditions in the 6 months before screening: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient cerebral ischemia Onset or symptomatic pulmonary embolism. Patients with known coronary artery disease, congestive heart failure that does not meet the above criteria or left ventricular ejection fraction <50% must adopt an optimized and stable medical plan determined by the treating doctor. If appropriate, you can consult a cardiologist.

  6. Received systemic anti-tumor therapy such as targeted therapy and biological drug therapy within 3 weeks before the first dose; Have received any Chinese herbal medicine or proprietary Chinese medicine with anti-tumor indications within 7 days before the first dose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 months
  the proportion of patients achieving the optimal overall remission (complete or partial remission)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | two year
  the time from the start of treatment to the first observation of disease progression or death from any cause (whichever occurs first)
Overall survival (OS) | two years
  the time from the start of treatment to death from any cause
Safety evaluation | two years
  NCI-CTCAE version 5.0 to assess adverse events (therapeutic toxicity)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xiaochang Gong, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No